CLINICAL TRIAL: NCT04031027
Title: DARWIN: Description of Apremilast Real World Italian Psoriasis Network - a Multicenter, Observational, Cross-sectional Study to Describe Patient Characteristics and Treatment Pattern
Brief Title: A Study to Describe the Characteristics of Patients Treated With Apremilast for Plaque Psoriasis in Italian Routine Clinical Practice
Acronym: DARWIN
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-026; U1111-1236-1175 (Other: WHO)
Record Dates: First submitted 2019-07-06; First posted 2019-07-24 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis
Keywords: apremilast; DARWIN; dermatology; retrospective; observational; psoriasis; cross-sectional
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Apremilast — Apremilast is prescribed in accordance with the terms of the SmPC and the marketing authorizations.
  Other Names: Otezla; CC-10004

SUMMARY:
The DARWIN study is an Italian multicenter, observational, cross-sectional study involving both a primary data collection (at enrollment visit) and secondary use of data (retrospective observation period). DARWIN will describe patients' characteristics in Italian routine clinical practice as well as the medication utilization patterns, including needs and benefits form the patient's perspective.

DETAILED DESCRIPTION:
The DARWIN study is anticipated to enroll 375 participants from 24 Italian dermatologic departments and recruitment is expected to take approximately 20 months. Participants must have started apremilast treatment 6 (±1) months prior enrollment in order to be considered eligible. The decision to prescribe apremilast falls within current practice according to the current decision-making process in the Italian routine clinical practice and according to AIFA prescribing information. No extra-procedures (diagnostic or monitoring) will be implemented and the assessment schedule reflects the routine clinical practice for psoriatic patients treated with apremilast. Patients will be consecutively enrolled in the study and information will be collected as recorded in the medical chart before starting apremilast (as close as possible to the apremilast start date/index date), and/or directly observed during the enrolment visit. The study variables will describe patient disease and characteristics, apremilast utilization patterns, psoriasis severity a, extent and impact on patient wellbeing, apremilast safety profile and apremilast satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Must have understood and voluntarily signed the informed consent and privacy form.
2. Age ≥ 18 years at the time of signing the informed consent and privacy form.
3. Patients with available hospital medical chart since the start of apremilast treatment ('index date').
4. Diagnosis of plaque psoriasis.
5. Treatment with apremilast for plaque psoriasis, according to Summary of Product Characteristics (SmPC), started 6 (±1) months before enrollment. Patients who interrupted apremilast treatment before enrollment will also be included.
6. Ability to understand (read & write) the Italian language and to follow the study instructions.

Exclusion Criteria:

1. Refusal to participate in this study or current participation in the treatment phase of an interventional clinical trial.
2. Started apremilast as part of a clinical trial, or previous apremilast use (prior to the index date).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patients ≥18 years
  * Moderate to severe plaque-type psoriasis according to Summary of Product Characteristics
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Mean age of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior enrolment)
  Age at treatment initiation (years)
Gender frequency of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Gender (male/female); frequency in %
Mean body weight of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Body weight in kg
Mean body mass index of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  BMI (combined outcome of weight and height in the form of kg/m^2)
Mean blood pressure of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Blood pressure in mmHg
Mean duration of psoriatic disease of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Duration in years
Mean Psoriasis area severity index score of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Psoriasis area severity index score (PASI)
Mean Body surface area of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Psoriasis-involved body surface area (BSA) in %
Mean Physician global assessment (PGA) score of the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Physician global assessment (PGA)
Frequency of previous antipsoriatic treatments in the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Previous treatments classes in %
Reasons for discontinuation of previous antipsoriatic treatments in the patients treated with apremilast | At treatment initiation (retrospective analysis, about 6 (+/-1) months prior prior enrolment)
  Frequency distribution of reasons in %

SECONDARY OUTCOMES:
Proportion of participants receiving apremilast at enrollment visit | Up to approximately 7 months after treatment initiation
  Persistence on apremilast treatment will be measured up to approximately 7 months after treatment initiation
Apremilast treatment duration | Up to approximately 7 months after treatment initiation
  Apremilast treatment duration is defined as the difference between the start date and the end date of apremilast treatment.
Change from baseline in Body Surface Area (BSA) | Up to approximately 7 months after treatment initiation
  BSA is measurement of the body area involved in relation to the whole body surface.
Change from baseline in the Physician Global Assessment (PGA) Score | Up to approximately 7 months after treatment initiation
  A 4 to 6-point scoring system used to assess plaque psoriasis disease severity
Change from baseline in the Dermatology Life Quality Index (DLQI) score | Up to approximately 7 months after treatment initiation
  DLQI is 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument.
Proportions of patients achieving PGA score 0 or 1 | Up to approximately 7 months after treatment initiation
  The Physician's Global Assessment is a measurement of overall involvement by the investigator at the time of evaluation. The sPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling, and plaque elevation. When making the assessment of overall severity, the investigator factored in areas that had already been cleared (ie, had scores of 0), not limited to the evaluation of remaining lesions for severity; consequently, the severity of each sign was averaged across all areas of involvement, including cleared lesions.
Proportions of patients achieving DLQI score ≤5 | Up to approximately 7 months after treatment initiation
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the subject is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Proportions of patients achieving ≥4 points improvement in DLQI score | Up to approximately 7 months after treatment initiation
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the subject is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Adverse Events (AEs) | Up to approximately 7 months after treatment initiation
  Descriptive analysis of AEs will be provided by severity, causality and seriousness
Treatment Satisfaction Questionnaire for Medication (TSQM) outcome score | Up to approximately 7 months after treatment initiation
  The TSQM-9 is a self-administrated instrument to understand a subject's satisfaction on the current therapy
Patient Benefit Index for Skin Diseases Score (standard version) (PBI-S) outcome score | Up to approximately 7 months after treatment initiation
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- Italy (16):
  - SOD Clinica Dermatologica A.O.U. Riuniti Umberto I Lancisi Salesi, Ancona, AN
  - UOC Dermatologia ASST Spedali Civili, Brescia, BS
  - Dermatologia Azienda Ospedaliera Papardo, Messina, ME
  - Dermatologica e Venereologia Univ. A.O.U. Consorziale Policlinico, Bari
  - UOS Clinica Dermatologica Ospedale San Giovanni di Dio, Cagliari
  - Dermatologia A.O.U. Policlinico-Vittorio Emanuele PO S.Marco, Catania
  - UOC Dermatologia Arcispedale Sant'Anna, Cona
  - Dermatologia Ospedale Piero Palagi, Florence
  - UOC Dermatologia A.O.U. Policlinico G. Martino, Messina
  - Dermatologia A.O.U. Federico II, Napoli
  - UOC Clinica Dermatologica A.O.U. Università della Campania Vanvitelli, Napoli
  - Dermatologia A.O.U. Maggiore della Carità, Novara
  - UOC Dermatologia e MST A.O.U. Policlinico P. Giaccone, Palermo
  - Clinica Dermatologica Policlinico Tor Vergata, Roma
  - Dermatologia e Venereologia A.O.U. Policlinico Umberto I, Roma
  - UOC Dermatologia Universitaria Ospedale A. Fiorini, Terracina

REFERENCES:
- [Background] Giofre C, Fabbrocini G, Potenza C, Tiberio R, Gisondi P, Marasca C, Nuzzo CMA, Benincasa E, Bianchi L; DARWIN study group. Real-World Apremilast Use for Treatment of Plaque Psoriasis in Italy: Patient Perspective, Characteristics, and Clinical Outcomes from the DARWIN Study. Adv Ther. 2023 Jul;40(7):3021-3037. doi: 10.1007/s12325-023-02516-y. Epub 2023 May 12. PMID 37171752
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com